CLINICAL TRIAL: NCT02043730
Title: A Phase II Randomized Trial Comparing a Combination of Abraxane and Gemcitabine Versus Gemcitabine Alone as First Line Treatment in Locally Advanced Unresectable Pancreatic Cancer. GAP (Gemcitabine Abraxane Pancreas) Trial
Brief Title: Abraxane and Gemcitabine Versus Gemcitabine Alone in Locally Advanced Unresectable Pancreatic Cancer.
Acronym: GAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Unità Sperimentazioni cliniche (Unknown); Istituto Nazionale Tumori di Napoli (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-002973-23
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer Stage II
Keywords: pancreatic cancer; locally advanced; unresectable cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- nab-paclitaxel and gemcitabine (Experimental): ARM A: nab-paclitaxel 125 mg/mq over 30 min and gemcitabine 1000 mg/mq weekly on days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Nab-paclitaxel and Gemcitabine; Drug: Gemcitabine
- Gemcitabine (Active Comparator): ARM B: Gemcitabine 1000 mg/mq over 30 minutes on days 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel and Gemcitabine — Chemotherapy will consist of nab-paclitaxel 125 mg/mq over 30 min and gemcitabine 1000 mg/mq weekly on days 1, 8 and 15 of a 28-day cycle
  Other Names: abraxane; gemzar
  Arms: nab-paclitaxel and gemcitabine
Drug: Gemcitabine — gemcitabine 1000 mg/mq over 30 minutes on days 1, 8 and 15 of a 28-day cycle.
  Other Names: gemzar

SUMMARY:
Pancreatic cancer is the fourth cause of cancer mortality: there are different treatment approaches to locally advanced pancreatic cancer management.

Generally, gemcitabine alone is considered a reasonable approach for advanced pancreatic cancer patients but we need a chemotherapeutic regimen able to prevent as much as possible a progression of the disease. Nab-paclitaxel (Abraxane) recently demonstrated an interesting activity profile in advanced pancreatic cancer. A combination of Nab-paclitaxel and gemcitabine has been demonstrated superior to gemcitabine alone in metastatic patients.

DETAILED DESCRIPTION:
Study population: Locally advanced unresectable pancreatic cancer patients

Elegibility criteria:

* Written informed consent
* Age >18 < 75 years
* Histologically/cytologically confirmed locally advanced, unresectable pancreatic cancer
* At least one lesion measurable with CT or MRI scan
* Performance Status (ECOG) 0-1 at study entry
* Life expectancy of at least 3 months
* Adequate marrow, liver and renal function
* Effective contraception if the risk of conception exists (in the Informed Consent for the patients the descriptions of possible contraceptives is reported

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >18 < 75 years
* Histologically/cytologically confirmed locally advanced, unresectable pancreatic cancer
* At least one lesion measurable with CT or MRI scan
* Performance Status (ECOG) 0-1 at study entry
* Life expectancy of at least 3 months
* Adequate marrow, liver and renal function
* Effective contraception if the risk of conception exists (in the Informed Consent for the patients the descriptions of possible contraceptives is reported)

Exclusion Criteria:

* Previous chemotherapy or radiotherapy for pancreatic cancer
* Severe cardiovascular disease
* Thrombotic or embolic events
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease
* Known hypersensitivity to study drug
* Known drugs or alcohol abuse
* Pregnant or breastfeeding women
* Previous or concurrent malignancy; except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and with evidence of no recurrence for at least 5 years prior to randomization
* Unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Progression Rate | progression rate is evaluated after 3 cycles of chemotherapy
  Assuming an expected progression rate in the control arm of 40% and an auspicated progression rate in the experimental arm of 20%,with one-tailed alpha=0.05, 80% power, 124 patients are required for the final analysis

SECONDARY OUTCOMES:
Quality of Response | Response to treatment is evaluated according to the RECIST criteria at the end of chemotherapy
  All patients must be considered in response analysis, including those who discontinue treatment or who die for any reason prior to response evaluations
Esplore the effects of nab-paclitaxel in terms of toxicity | every 3 cycles of chemotherapy
  Treatment-emergent adverse events, drug-related adverse events and safety laboratory parameters will be analysed by treatment groups and CTCAE grade
Progression Free Survival | time from the start of the treatment until PD or death
  Progression free survival time will be defined as the time from randomization until the date of first observed disease progression (radiological or clinical, whichever is earlier) or death due to any cause, if death occurs before progression is documented.
  Patients who did not progress will be censored at the last date they were known to be alive.
  Patients who died of disease and for whom a date of progression is not available will be considered to have progressed on the day of their death
Overall Survival | the time from randomization to the date of death
  Overall survival time will be defined as the time from randomization to the date of death. If the subject has not died, survival will be censored on the last date the subject was known to be alive (last date of follow up).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cascinu, PhD, Study Chair — GISCAD Foundation
Locations (39):
- Italy (39):
  - A.O. Universitaria Ospedali Riuniti, Ancona, AN
  - Istituto Tumori Giovanni Paolo II, Bari, BA
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - A.O. Humanitas Gavazzeni, Bergamo, BG
  - A.O. Ospedale G.Rummo, Benevento, BN
  - ASDAA Bolzano, Bolzano, BZ
  - Policlinico Universitario D.Casula, Monserrato, Cagliari
  - Azienda Ospedaliera Sant'Anna, Como, CO
  - A.O. Ospedale S.Martino, Genova, GE
  - A.O. Polo Oncologico Vito Fazzi, Lecce, LE
  - Azienda Ospedaliera San Gerardo di Monza,, Monza, MB
  - Ospedale Civile, Legnano, MI
  - Azienda Ospedaliera San Paolo, Milan, MI
  - Policlinico, Modena, MO
  - AUSL di Piacenza, Piacenza, PC
  - ULSS15 di Camposampiero/Cittadella, Camposampiero, PD
  - Ospedale Santa Croce, Fano, Pesaro
  - Azienda Ospedaluiera Universitaria, Parma, PR
  - A.O. S.Salvatore, Pesaro, PS
  - IRCCS F.S. Maugeri, Pavia, PV
  - Ospedale Civile, Vigevano, PV
  - Azienda Ospedaliera Ospedale San Carlo, Potenza, PZ
  - Ospedale Civile degli Infermi, Faenza, Ravenna
  - Ospedale Umberto I, Lugo, Ravenna
  - Azienda Ospedaliera, Ravenna, RA
  - A.O. S.Maria Nuova - IRCCS, Reggio Emilia, RE
  - Azienda Policlinico Umberto I, Roma, RM
  - A.O. Cà Foncello, Treviso, TV
  - Ospedale di Circolo, Busto Arsizio, Varese
  - AO Papa Giovanni XXIII, Bergamo
  - Ospedale degli Infermi, Biella
  - Casa di Cura di Poliambulanza, Via Bissolati 57, Brescia
  - A.O. Careggi-Università, Viale Pieraccini, 17, Florence
  - AOU Policlinico Universitario Federico II, Napoli
  - INT-IRCCS Fondazione G.Pascale, Napoli
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Policlinico Universitario A.Gemelli, Roma
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma
  - Ospedale di Sondrio, Sondrio

REFERENCES:
- [Derived] Cascinu S, Berardi R, Bianco R, Bilancia D, Zaniboni A, Ferrari D, Mosconi S, Spallanzani A, Cavanna L, Leo S, Negri F, Beretta GD, Sobrero A, Banzi M, Morabito A, Bittoni A, Marciano R, Ferrara D, Noventa S, Piccirillo MC, Labianca R, Mosconi C, Casadei Gardini A, Gallo C, Perrone F. Nab-paclitaxel/gemcitabine combination is more effective than gemcitabine alone in locally advanced, unresectable pancreatic cancer - A GISCAD phase II randomized trial. Eur J Cancer. 2021 May;148:422-429. doi: 10.1016/j.ejca.2021.02.023. Epub 2021 Mar 31. PMID 33812334